CLINICAL TRIAL: NCT02330016
Title: Juvederm Voluma® XC for the Treatment of Hypoplastic Chin
Acronym: VolumaChin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kenneth Beer (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Kenneth Beer, President, Beer, Kenneth R., M.D., PA
Organization: Beer, Kenneth R., M.D., PA (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VolumaChin-001
Record Dates: First submitted 2014-12-17; First posted 2015-01-01 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Mandibular Hypoplasia
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voluma XC (Experimental): Injections of Voluma will be accomplished using a serial puncture and fanning technique with the needle inserted to the periosteal plane as well as in the subcutaneous plane. The treatment area will include the medial and lateral chin as defined: lateral chin landmark is the depressor anguli oris.
  Interventions: Device: Voluma XC

INTERVENTIONS:
Device: Voluma XC — Voluma XC

SUMMARY:
This is a single center study of the safety and efficacy of Juvedérm Voluma for the treatment of hypognathism.

Each qualified subject will undergo treatment with Juvedérm Voluma in the anterior and lateral chin for volume correction. Prior to treatment, the principal investigator will evaluate the severity of chin recession using a 90 degree image and a goniometer to measure the angle from the glabella to the chin. Subjects will be eligible for injection if the angle measures between 145 - 160 degrees. Facial digital photography will be captured prior to treatment and at each subsequent visit. The subject will complete a safety and injection site response (ISR) diary beginning on the evening of treatment.

The subject will return at Day 3 and Day 14 after initial treatment, at which time the subject will undergo photography and the investigator will rate treatment improvement (GAIS). An independent image analysis technician will assess the degree of correction. The investigator will evaluate the treatment area for any adverse events (AEs).

The subject will return 30 days after initial treatment, and the principal investigator will determine if a touch-up treatment is warranted. If deemed necessary, a touch-up treatment may be administered. Facial digital photography will be captured prior to treatment and following treatment. The subject will return 3 days after the touch-up to undergo digital photography and for the principal investigator to assess safety/improvement.

After initial or touch-up treatment, whichever is last, routine follow-up visits for safety and effectiveness will occur at 1 (30 days), 2, 4, 6, 9 (telephone call only) and 12 months. At all follow-up visits, facial digital photography will be captured and the investigator will rate treatment improvement (GAIS).. At screening and at Months 1, 2, 4, 6 and month 12 subjects will complete the satisfaction of face overall module of the FACE-Q questionnaire.

The goal of this study will be to assess the feasibility of Voluma XC for the treatment of hypoplastic chins

DETAILED DESCRIPTION:
Primary Objective: To evaluate efficacy of Voluma XC for the treatment of hypoplastic chins.

Secondary Objective: To evaluate patient satisfaction and improvement of GAIS following treatment with Voluma for hypoplastic chins.

The expected outcome following deep (dermal and/or supra periosteal) injection of Voluma when used to treat hypognathism is significant improvement in the facial angle of the chin. Significant improvement defined as the mean change in the facial angle of the face measured by the blinded digital image analysis technician. A secondary effectiveness measure will be patient and treating investigator measure of improvement using the FACE-Q questionnaires as well as the mean change in the GAIS score.

The study will span a total of approximately 15 months: an estimated 2 months for recruitment and 12 months for follow-up. Each subject's participation will encompass a screening/baseline visit, Day 3 and a Day 14 visit with a possible 1 month touch up (if touch up occurs then a day 3 and a day 14 and a month 1 will occur following the touch up then followed by study visits at 2, 4, 6, month and a 9 month telephone safety visit and a 12 month clinic visit (end of study).

JUVÉDERM® Voluma XC Injectable Gel No control treatment will be used. The primary effectiveness endpoint will be one month after optimal correction has been attained according to the investigator.

The image analysis technician performing the evaluation will be blinded as to the amount of product injected. All digital photos will be analyzed in a batched, randomized format (including the pre-treatment photos) in order to blind the technician.

Retreatment Criteria (if applicable) Study subjects will return for possible touch up 1 month following initial injection. At this time, the investigator and the subject will evaluate the outcome of the initial treatment. In the event that both the subject and the investigator concur that additional treatment is indicated because of a suboptimal aesthetic correction, a repeat injection of Voluma XC will be performed. If a repeat treatment does take place then the subject will then be followed at Day 3 and Day 14 and Day 30. In the event that the subject does not want retreatment the subject will remain in the study and followed through the course of the trial.

The subject will undergo treatment and return for follow-up visits throughout the study period. At each visit, the Principal Investigator or designee will record AEs and concomitant medications, therapies, and treatments. All reported AEs will be documented. The procedures to be performed at each visit are described below.

Injections of Voluma will be accomplished using a serial puncture and fanning technique with the needle inserted to the periosteal plane as well as in the subcutaneous plane. The treatment area will include the medial and lateral chin as defined: lateral chin landmark is the depressor anguli oris.

Photography will be mandatory to participate in this clinical trial. Subjects will consent to allow Kenneth R. Beer, M.D., PA permission to use photographs for FDA advisory panel meetings, scientific journals and conferences, advertising, publicity, and promotional purposes as one option. Additional options will be given to the subject to allow Kenneth R. Beer, M.D., PA to only use photographs for FDA advisory panel meetings and scientific journals and conference, but does NOT have permission to use the photographs for advertising, publicity, or promotional purposes as option 2. The third and final option allows the subject to have photographs taken, but subject does NOT give permission to use photographs for FDA advisory panel meetings, scientific journals and conferences, advertising, publicity, and promotional purposes.

The photographs will be taken with 3D photography system and will be analyzed by a third party which is hired by the sponsor. Full confidentiality cannot be maintained due to the entire face will be photographed. Confidentiality will try to be maintained by only using subject identifiers. If at a later date the subject does not want photos used for other purposes that were consented to the subject at any time during the course of the study will be allowed to change and update the photograph consent. If subject withdraws all photo consent the subject will be discontinued from the study since photographs are mandatory to participate in this clinical study.

The Principal Investigator will ensure that each subject meets the eligibility criteria. The Principal Investigator will capture a 90 degree angle photo and using a goniometer to manually measure the angle between the glabella and the mentalis and subjects with angles between 145-160° will be included in the study. The Principal Investigator or designee will record reasons for those subjects who withdraw consent prior to randomization or who do not meet the inclusion/exclusion criteria.

The Principal Investigator or designee will collect and record the subject's demographic information, medical and surgical history, cosmetic procedures history, and Fitzpatrick skin phototype.

Initial Treatment Visit (Day 0) If Screening and Day 0 visit are on the same day, all procedures performed at Screening will be performed at Screening will be performed once, prior to treatment administration.

Prior to treatment, vital signs (blood pressure, heart rate, respiration rate, and temperature only) will be measured. Study staff will attain subject demographics, medical, cosmetic, and dental history. A negative UPT test will be confirmed prior to randomization. Photos will be taken with the Canfield Vectra 3D system. Subjects will be asked to complete the FACE-Q questionnaire licensed by Memorial Sloan Kettering (3). Concomitant medications will be captured. A subject diary will be given to each subject to complete for 30 days. A Investigator assessment of chin function will be completed prior to injections.

Day 3 (+/- 2days) Subject will return to clinic for Day 3 follow up. Subject will be photographed with the Canfield Vectra 3D system and the investigator will rate the improvement using the GAIS score and Investigator Assessment of chin function.

Day 14 (+/-3 days) Subject will return to clinic for Day 14 follow up. Subject will be photographed with the Canfield Vectra 3D system and the investigator will rate the improvement using the GAIS score and Investigator Assessment of chin function.

Day 30 retreatment visit or Month 1 visit (+/-7days) Subject will be assessed by investigator to determine if retreatment is needed. If no retreatment occurs then visit will become the one month visit.

Month 1 Visit Subject will be photographed with the Canfield Vectra 3D system, investigator GAIS score and FACE Q questionnaire completed, adverse events captured, collection of diary, and concurrent procedures documented.

Retreatment Visit If retreatment is needed the visit schedule will be as follows from the date of retreatment day 3 (+/- 2 days), day 14 (+/- 3 days) and then day 30 (+/- 7 days). Subject and investigator will then complete Month 1 visit requirements as documented above. (Same procedures will be followed from initial injection) Month 2 (+/- 14 days) Subject will be photographed with the Canfield Vectra 3D system, investigator GAIS score, and Investigator Assessment of chin function, Face Q questionnaire, adverse events and concurrent procedures captured.

Month 4 (+/- 14 days) Subject will be photographed with the Canfield Vectra 3D system, investigator GAIS score, and Investigator Assessment of chin function, Face Q questionnaire, adverse events and concurrent procedures captured.

Month 6(+/- 14 days) Subject will be photographed with the Canfield Vectra 3D system, investigator GAIS score, and Investigator Assessment of chin function, Face Q questionnaire, adverse events and concurrent procedures captured.

Month 9 (+/- 14 days) telephone safety call Subject will be called to review any new concomitant medications or any new adverse events since month 6 visit.

10 Month 12 (+/-14 days) End of Study Visit Subject will be photographed with the Canfield Vectra 3D system, investigator GAIS score, and Investigator Assessment of chin function, Face Q questionnaire, adverse events and concurrent procedures captured. End of Study page completed Instructions for the Subjects

* Following injection with Voluma, application of ice for 10 minutes per hour while awake may help to reduce swelling and this may be used for a period of 3-5 days.
* Discomfort may be treated with acetaminophen.
* Gentle massage may also be used to minimize lumps and bumps which are more common during the first 7 days following treatment.

ELIGIBILITY:
Inclusion Criteria:

Male or female, 22 years and above Has moderate to severe chin hypognathism Moderate to severe hypognathism 145-160 degrees as measured with goniometer by principal investigator at screening visit. All other measurements will be performed by a blinded Canfield facial image analysis technician. Written informed consent has been obtained Written Authorization for Use and Release of Health and Research Study Information has been obtained Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable. Ability to follow study instructions and likely to complete all required visits If the subject is a female of childbearing potential (sexually active and not sterile, surgically sterilized, or postmenopausal with no menses for at least 1 year), have a urine pregnancy test evaluated as negative at randomization, have used contraception for at least 30 days prior to enrollment, and agree to use a reliable method of contraception for the duration of the study. Subject agrees to abstain from any treatment to the lower 1/3 of the face including botulinum toxins, hyaluronic acid fillers, cosmetic surgery, laser/light therapy, chemical peels, etc.

Exclusion Criteria:

Uncontrolled systemic disease. Severe cardiovascular disease. Known allergy or sensitivity to the study medication(s) or its components Females who are pregnant, nursing, or planning a pregnancy. Pregnancies that occur will be followed by the sponsor until delivery or termination. Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study and for the duration of the study. Previous treatment to the glabella, philtrum or chin with hyaluronic acid fillers or semi-permanent filler (i.e. Radiesse) in the past 12 months and for the duration of the study Any use of permanent filler materials such as Artefill or silicone in the face. Subjects planning a facial cosmetic procedure during the study period or with prior cosmetic procedures (i.e. surgery) in the treatment area or visible scars that may affect the evaluation.

Subjects will need to be on the same facial product regimen for 90 days and no topical anti-wrinkle products on the chin. Had received (or was planning to receive) anti-coagulation medication(e.g., warfarin) from 10 days pre to 3 days post-injection. Planned rhinoplasty Any subjects with volume deficit due to trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disese, or HIV-related disease. Infection or dermatoses at the injection site.

Evidence of recent alcohol or drug abuse. Medical and/or psychiatric problems that is severe enough to interfere with the study results.

Known bleeding disorder or is receiving medication that will likely increase the risk of bleeding as the result of injection. Has facial hair that would interfere with evaluation and treatment of the chin area Has a tendency to develop hypertrophic scarring Has a history of anaphylaxis or allergy to lidocaine (or any amide-based anesthestics), HA products, or Streptococcal protein.

Has porphyria Has an active inflammation, infection, cancerous or precancerous lesion, or unhealed wound in the lower face/jawline or chin area.

Subject has a condition or is in a situation which in the Investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Primary outcome will be a change in the facial angle as measured by a blinded facial image analysis technician. | 12 months

SECONDARY OUTCOMES:
Evaluation of the patient's self image using the satisfaction with lower face and jawline, satisfaction of chin, and appraisal of area under chin modules of the FACE-Q questionnaire. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Beer, M.D., Principal Investigator — Beer, Kenneth R., M.D., PA
Locations (1):
- Kenneth R. Beer, M.D., PA, West Palm Beach, Florida, United States

REFERENCES:
- See also: practice webste — http://palmbeachcosmetic.com